CLINICAL TRIAL: NCT05456776
Title: Azathioprine Linked With Impaired Intestinal Epithelial Postoperative Regeneration in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: nr 2803/2012
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: azathioprine, immunomodulators; epithelial repair; restitution, regeneration; cellular damage; Crohn's disease; apoptosis, p53, caspase-3, Ki67
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Intestinal samples from macroscopically healthy margins of surgical specimens. Two, one-centimeter each, fragments of the small intestine were cut off from the proximal end of the specimen (S1, S2) and analogous two from the large intestine (L1, L2) of the distal end. Then, all samples were inherently prepared and transferred for immunofluorescence (S1, L1) and Western-blot (S2, L2) analysis, while the whole remaining specimen delivered for histopathological examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
What is known?

* the impact of AZA, immunomodulatory drug widely used in active CD, on the intestinal wall differs from those of steroids, what is reflected in the significant difference in the postoperative anastomotic leaks rate
* AZA inhibits intestinal epithelial cell growth by inducing the apoptosis and inhibiting proliferation of intestinal epithelial cells in in vitro studies What is new?
* The effect of AZA on cellular damage was assessed in humans' study
* AZA increases cell apoptosis in the intestinal epithelium of active CD patients, much stronger than steroids
* AZA actively promotes the DNA damage repair in the intestinal epithelium; the steroid effect, even when combined with AZA, is not so pronounced
* The intensity of proliferative processes, in contrast to steroids, is significantly inhibited in response to AZA
* The disintegration of the mucosa layer in response to AZA is observed
* The difference in the mechanisms of action of AZA and steroids on the intestinal mucosa may be directly related to the reported difference in the risk of septic postoperative complications, but this requires further research

DETAILED DESCRIPTION:
Although conservative treatment of Crohn's disease (CD) is constantly improving some patients still require surgery. Optimal perioperative management includes pharmacological modifications to reduce complications risk. Unfavorable effect of steroids and from recently also biologics on intraabdominal and wound septic complications is known, but until now azathioprine (AZA) is considered to be safe.

The aim of our study was to assess the impact of AZA on intestinal epithelial cells damage as well as restoration and regeneration in patients with active CD as a surrogate marker of healing. We assessed intestinal specimens taken from macroscopically healthy surgical margins of all consecutive CD patients operated due to active isolated ileocecal disease during the study period (2014-2016) in tertiary referral center. We immunohistochemically tested expression of Ki-67, caspase-3 and p-53 as a markers of cell proliferation, apoptosis and DNA damage respectively. Quantitative evaluation of cellular expression of determined proteins was assessed using a confocal microscope. We also performed immunofluorescent tests for cellular integrity using ZO-1 and E-cadherin proteins expression. Additionally we assessed 30 days clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with histopathologically confirmed CD at least six months earlier, operated due to active disease characterised by clinical, endoscopical, and radiological findings
* ileocecal involvement
* No other CD manifestations
* Signed informed consent

Exclusion Criteria:

* Previous bowel surgery for CD
* Presence of severe, progressive, uncontrolled cardiological, pulmonary, nephrology, contagious or psychiatric illness whose course could affect the patient's risk of perioperative complications
* Significant disease symptoms so far undiagnosed
* Present or suspected malignancy or previous oncological treatment in the last five years
* Cardiac stimulator or cardioverter-defibrillator
* Pregnancy
* Severe non-abdominal surgery or severe trauma in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The eligible population were male and female patients diagnosed with histopathologically confirmed CD at least six months earlier, operated due to active disease characterised by clinical, endoscopical, and radiological findings. Qualification to surgery was performed by multidisciplinary team consisting of surgeon, gastroenterologist, endoscopist and radiologist and was based on those data. Only patients with isolated ileocecal involvement were included for further evaluation.
  For the purpose of the study, we divided our cohort into four groups accordingly to preoperative treatment: group N - patients treated with no immunomodulators, group S - patients on steroids, group A - patients on AZA, and group AS - on combination therapy (AZA + steroids).
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
histopathological assessment of the azathioprine's impact on intestinal damage | 30 days
  Comparison of the impact of immunomodulatory drugs on regeneration and restoration of small and large bowel's epithelial cells not affected by Crohn's disease.
  It was immunohistochemical assessment of expression of caspase-3, p-53 and Ki-67 as a markers of cell apoptosis, DNA damage and proliferation, respectively. But all of those stainings were then assessed by histopathologist in white light microscope.
  Quantitative evaluation (counting in high power field) of cellular expression of determined proteins was assessed using a confocal microscope.